CLINICAL TRIAL: NCT06279169
Title: The Effect of Heart Sound and White Noise on Pain and Physiological Parameters During Hepatitis B Vaccine Injection in Newborns: A Randomized Controlled Trial
Brief Title: The Effect of Heart Sound and White Noise on Pain and Physiological Parameters During Hepatitis B Vaccine Injection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bartın Unıversity (Other)
Responsible Party: Principal Investigator, Fatma Dinç, Principal Investigator, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-BRT-SBF-113355
Record Dates: First submitted 2024-02-17; First posted 2024-02-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Pain, Acute; Newborn; Vitality
Keywords: Pain; Acute Pain
MeSH Terms: conditions — Acute Pain; Pain | interventions — Heart Sounds

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heart sound group (Experimental): In the heart sound group, the heart sound with an average heart rate of 70 beats is transmitted to the loudspeaker via an Mp3 player. Two small 200 W loudspeakers (SONY®)/"JBL" brand loudspeakers are used, placed on either side of the newborn's head, 30 cm from the newborn's ears.
  Interventions: Behavioral: Heart Sound
- White noise group (Experimental): In the white noise group, the mother of the baby is told that the white noise to be used in the study will be used for pain relief. For the white noise, the musician Osman Orhan's colic album, which was released by the production and often used in the literature. The song "Bebeğiniz Ağlamasın Pt-3" from the album "Kolik" will be used (permission to use it in this work has been granted by ON Music Production). The volume is set to 45 db. The "JBL" loudspeaker is placed on the newborn's toe 5 minutes before the procedure, about 30 cm from the newborn's ear, and white noise is played 5 minutes before, during (at the 1st minute) and 5 minutes after the administration of the Hep B vaccine.
  Interventions: Behavioral: White Noise
- Control (No Intervention): Newborns in the control group will not receive any intervention other than Hepatitis B vaccination.

INTERVENTIONS:
Behavioral: Heart Sound — In the Heart sound group, this sound will be played to the newborn 5 minutes before Hep B vaccine administration, during the procedure (at 1 minute) and 5 minutes after Hep B vaccine administration
  Arms: Heart sound group
Behavioral: White Noise — Musician Osman Orhan's song "Bebeğiniz Ağlamasın" from his album Kolik will be used for white noise. The volume will be set to 45 db.
  Arms: White noise group

SUMMARY:
It can cause physiological and behavioral changes in infants such as pain, tachycardia, hypoxemia, increased blood pressure, grimacing, prolonged crying, and irritability. Vaccination is an important part of neonatal nursing care. Newborns express their pain nonverbally and behaviorally. Therefore, any pain assessment is based on the ability of others to recognize pain symptoms. This randomized controlled trial was planned to evaluate the effect of heart sound and white noise on pain and physiological parameters during intramuscular injection of hepatitis B vaccine in newborns. This randomized controlled study used parallel trial design.

DETAILED DESCRIPTION:
The research hypotheses are H1: Neonates in the heart sound group will have lower procedural pain scores than neonates in the control group. H2: Neonates in the white noise group will have lower procedural pain scores than neonates in the control group. H3: Neonates in the heart sound group have lower procedural heart rate peak values than neonates in the control group. H4: Neonates in the white noise group have lower procedure-related peak heart rates than neonates in the control group. H5: Neonates in the heart sound group have higher procedural oxygen saturation values than neonates in the control group. H6: Neonates in the white noise group have higher procedural oxygen saturation values than neonates in the control group.

Methods The study was designed as a randomized controlled trial. The population of this study will consist of newborns who are followed up at Bartın Maternity and Children's Hospital. Statistical power, type I error, effect size, and study design will be taken into account when calculating the sample size. The study will be designed to have a power of at least 80% and a type I error rate of 5%. As there is no similar study evaluating the effect of heart tones and white noise on pain and physiological parameters during hepatitis B vaccination in children, the effect size of the study will be aimed at medium (0.25) to determine the sample size. Based on a medium effect size (f: 0.25), 80% (1 - β error) power and 95% (α error) confidence level, and taking into account data loss, it was calculated that the sample size should be increased by 10%, and the sample size of 33 newborns in each group should consist of 99 newborns in total G*Power 3.1.9.7.

Before starting the study, mothers will be informed about the purpose of the study and the heart sound and white noise applications to be applied and their written informed consent will be obtained. After written informed consent has been obtained from the mothers, the newborns will be randomised to 3 groups (heart sound, white noise, control group) by a statistician independent of the study (www. randomize.org) using a computer program. All newborns will receive a standardised approach. Standardised approach: All Hep B vaccine administration will be performed by a nurse during the morning shift and administered intramuscularly through the vastus lateralis muscle at a 90-degree angle using a 1-inch 23-gauge needle to infants in all three groups. All conditions such as room temperature (25°C), light, injection procedure will be the same in all three groups. Neonates will be fed at least 30 minutes before the procedure. Care will be taken to avoid non-nutritive sucking, touching or swaddling the baby during the procedure to avoid confusion with other pain relief methods. Aseptic techniques are observed during all procedures.

During the implementation of the measurement tools, the researcher will go to the relevant facility herself and the data collection forms will be applied face to face. The researcher and the nurse will not use any aromatic substances in the baby monitoring room during the study.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 38-41 weeks,
* Newborn birth weight >2500 g
* Stable vital signs before the procedure,
* Postanatal age between 2-28 days,
* No contraindications to the administration of hepatitis B vaccine
* Delivery of the newborn to the mother after birth
* Consent of the parents of the newborn to participate in the study
* Fasting less than 3 hours/30 minutes before feeding
* A valid score on the newborn hearing screening test
* Newborn not crying before vaccination

Exclusion Criteria:

* Newborn babies requiring respiratory support,
* Newborns with any neurological disorder (seizures)
* Newborns taking opiates or born to mothers taking opiates
* Newborns receiving muscle relaxants, sedatives, analgesics
* Babies with major congenital anomalies
* Neonates with an APGAR score of less than 7 at 5 minutes
* Neonates who have undergone surgery
* Newborns with birth trauma (especially rapid delivery)
* Conditions that may prevent communication with parents (e.g. speech problem)
* Hearing impairment
* Newborns who will be transferred to another hospital

Ages: 2 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-08-29 (Estimated); Study Completion 2025-08-29 (Estimated)

PRIMARY OUTCOMES:
The Newborn Infant Pain Scale (NIPS) | 15 minutes
  Used to assess behavioral and physiological pain responses of preterm and term infants. The Neonatal Infant Pain Scale is a Likert-type scale consisting of 6 parameters including facial movements (0; relaxed, 1; restless), crying (0; no crying, 1; moaning, 2; loud crying), breathing (0; relaxed, 1; variable-irregular), arm (0; relaxed-free, 1; flexion-extension), leg (0; relaxed-free, 1; flexion-extension) and sleep-wakefulness (0; sleep-wakefulness peaceful, 1; restless). According to the scale, 7 is interpreted as the highest level of pain and 0 as the lowest level of pain. A high score indicates greater severity of pain.

SECONDARY OUTCOMES:
oxygen saturation | 15 minutes
  In each group, oxygen saturation of the newborns to be included in the study will be performed by the same researcher with the same calibrated pulseoximeter device in the infant monitoring unit.
heart rate | 15 minutes
  The heart rate measurements of the newborns to be included in the study in each group will be performed by the same researcher with the same calibrated device in the infant monitoring unit.
Crying Time | 15 minutes
  During the Hep B vaccination procedure, a stopwatch will be started from the moment the newborn starts crying. "Samsung" brand "Note 10" model phone stopwatch will be used for the stopwatch. During the procedure, the stopwatch will be turned on when the baby cries, and the stopwatch will be stopped when the crying stops.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No